CLINICAL TRIAL: NCT03071796
Title: Influence of Liquid Multivitamin Supplementation on Life Quality, Mood, Perception of Stress and Health-related Vital and Blood Parameters and the Immune System
Brief Title: Influences of Multivitamin Supplementation on Health Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Kuno Hottenrott, Prof., Prof. Dr.; University of Halle-Wittenberg, Department of Sports, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ILUG-201701
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multivitamin supplement (Experimental): liquid multivitamin supplement for 12 weeks
  Interventions: Dietary Supplement: multivitamin supplement
- placebo (Placebo Comparator): liquids with similar appearance and taste like multivitamin supplement for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: multivitamin supplement — supplement includes 97 natural extracts
  Arms: multivitamin supplement
Dietary Supplement: Placebo — liquids with similar appearance and taste like multivitamin supplement for 12 weeks
  Arms: placebo

SUMMARY:
In this study the investigator will evaluate whether a liquid multivitamin supplement influences blood and vital parameters. Furthermore the investigator will establish the effects on life quality, mood and perception of stress and will characterize changes on immune system.

DETAILED DESCRIPTION:
The double-blind, randomized intervention study is conducted for 12 weeks and includes two groups (placebo versus verum) with same number of participants.

The investigator aims to determine the effects of multivitamin supplement on blood and vital parameters which includes blood pressure, pulse, heart rate, variability of heart rate, vitamin D, vitamin B12, folic acid, homocysteine, HbA1c. Furthermore the investigator will access life quality, mood and perception of stress through the following questionnaire POMS, PSS-10, SF12 & SF36. The investigator will evaluate whether the multivitamin supplement changes the frequency of diseases like cold which represents the function of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* healthy women and men
* age between 30-60 years
* employed

Exclusion Criteria:

* acute and chronic diseases (including diabetes, inflammatory bowel diseases, dementia, multiple sclerosis)
* frequent use of alcohol, drugs or cigarettes (>5 cigarettes / day)
* use of additional supplements
* use of medications (e.g. antihypertensive medications, lipid reducers, thyroid medication)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Vitamin B12 | change measures (baseline to 12 weeks)
  vitamin B12 [pmol/l]

SECONDARY OUTCOMES:
Analysis of blood pressure | change measures (baseline to 12 weeks)
  blood pressure
Analysis of heart rate variability | change measures (baseline to 12 weeks)
  heart rate variability
Analysis of speed of pulse wave, | change measures (baseline to 12 weeks)
  speed of pulse wave
Plasma concentration of 25-hydroxyvitamin D | change measures (baseline to 12 weeks)
  25-hydroxyvitamin D [nmol/l]
Plasma concentration of folic acid | change measures (baseline to 12 weeks)
  folic acid [nmol/l]
Plasma concentration of homocysteine | change measures (baseline to 12 weeks)
  homocysteine [µmol/l]
Plasma concentration of HbA1c | change measures (baseline to 12 weeks)
  HbA1c [mmol]

OTHER OUTCOMES:
Susceptibility to infections | up to 12 weeks
  Documentation of diseases in disease diary
assessment of life quality | change measures (baseline to 12 weeks)
  use of questionnaires SF-36
assessment of mood | change measures (baseline to 12 weeks)
  use of questionnaires POMS
assessment of perceived stress | change measures (baseline to 12 weeks)
  use of questionnaires PSS-10

CONTACTS AND LOCATIONS:
Overall Officials: Kuno Hottenrott, Prof. Dr., Principal Investigator — University of Halle-Wittenberg, Department of Sports
Locations (1):
- University of Halle-Wittenberg, Halle, Germany

IPD SHARING:
Plan to Share IPD: No